CLINICAL TRIAL: NCT01800032
Title: Pilot Study of [18F] Fluorodeoxyglucose Positron Emission Tomography- Magnetic Resonance Imaging (FDG-PET-MRI) in CNS and Extra-CNS Tumors of Patients With Neurofibromatosis-1 (NF1)
Brief Title: PET/MRI in CNS and Extra-CNS Tumors of Patients With Neurofibromatosis-1 (NF1)
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC1222
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Neurofibromatosis-1; Optic Glioma; Plexiform Neurofibroma
MeSH Terms: conditions — Optic Nerve Glioma; Neurofibroma, Plexiform

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Plexiform Neurofibroma: NF1 associated plexiform neurofibroma
- Optic Glioma: NF1 associated optic glioma

SUMMARY:
This prospective pilot study is designed to provide preliminary data on the use of Fluorodeoxyglucose Positron Emission Tomography-Magnetic Resonance Imaging (FDG-PET-MRI) in patients with neurofibromatosis-1 (NF1) associated optic glioma and plexiform neurofibroma (PN).

Subjects will undergo FDG-PET-MRI scans in place of standard of care imaging at 0 and 12 months, unless more frequent imaging is clinically indicated. Subjects and their family caregivers will also undergo serial interviews and complete questionnaires related to the psychosocial aspects of NF1.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with neurofibromatosis-1 with either optic glioma, due for imaging scan, or plexiform neurofibroma, due for imaging secondary to clinical signs or symptoms of progressive disease
* ≥ 6 years of age
* English-speaking
* If female of child-bearing potential, negative urine pregnancy test performed within 7 days prior to each FDG-PET-MRI
* Study-specific informed consent or assent obtained and signed

Exclusion Criteria:

* Unable to undergo FDG-PET-MRI without sedation
* Currently undergoing chemotherapy for progressing optic glioma
* Pregnant or lactating female
* Poorly controlled diabetes mellitus
* Presence of pacemaker, intracranial aneurysm clip, cochlear implant, metal halo device, epicardial pacemaker leads, or any other device that makes MRI unsafe
* Serum creatinine > 1.8 mg/dL OR GFR < 30 mL/min
* Unable to lie flat for > 1 hour
* Body Mass Index (BMI) > 35

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: UNC Hospitals
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01-16 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2019-12-05 (Actual)

PRIMARY OUTCOMES:
Plexiform Neurofibroma Cohort: Difference in FDG-avidity between progressive and non-progressive lesions | 12 months
  Ratios of SUVmax values within a group of patients who all have progressive disease
Optic Glioma Patients: Compare FDG-avidity between patients with progressive and non-progressive disease | 12 months

SECONDARY OUTCOMES:
Report descriptive statistics for FDG-PET-MRI results | 0, 12 months
  SUV max, tumor/brain uptake ratio, tumor/muscle uptake ratio
Explore impact of FDG-PET-MRI surveillance on patient and family caregiver uncertainty and psychological distress | 0, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Gershon, MD, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina-Chapel Hill, Chapel Hill, North Carolina, United States